CLINICAL TRIAL: NCT00305942
Title: A Phase II Trial of Topotecan and Carboplatin in the First-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Topotecan and Carboplatin in the First-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 117
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Small Cell
Keywords: Lung Cancer; Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms | interventions — Topotecan; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Topotecan 4mg/m2 IV on days 1, 8.
  Carboplatin AUC=5 IV day 1 only .
  - Cycles are repeated every 21 days for > 4 cycles of topotecan and carboplatin (maximum 6 courses). Restaging studies will be performed every 2 cycles (or 6 weeks.)
  Interventions: Drug: Topotecan; Drug: carboplatin

INTERVENTIONS:
Drug: Topotecan — Topotecan 4mg/m2 IV on days 1, 8.
  Other Names: Hycamtin
Drug: carboplatin — Carboplatin AUC=5 IV day 1 only .
  Other Names: 41575-94-4

SUMMARY:
This proposed phase II trial will investigate the combination of topotecan/carboplatin in the first-line treatment of patients with extensive-stage SCLC. Topotecan/platinum regimens are emerging as common treatments for patients with extensive-stage disease. This trial will be one of the first clinical trials to evaluate a combination of weekly topotecan and carboplatin in the first-line treatment of extensive-stage SCLC.

DETAILED DESCRIPTION:
Eligible patients will receive treatment with carboplatin and topotecan.

Topotecan 4mg/m2 IV on days 1, 8.

Carboplatin AUC=5 IV day 1 only .

- Cycles are repeated every 21 days for > 4 cycles of topotecan and carboplatin (maximum 6 courses). Restaging studies will be performed every 2 cycles (or 6 weeks.)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed small cell lung cancer with extensive stage disease. This includes patients with stage IIIB and IV disease.
* Patients with small cell histology are eligible. Large neuroendocrine or mixed small cell and non-small cell histology are not eligible.
* Patients must have measurable or evaluable disease.
* ECOG performance status 0 or 1.
* Patients must have adequate bone marrow, liver and kidney function
* The patients may have had no previous chemotherapy.
* Patients must be able to understand the nature of the study and give written informed consent.

Exclusion Criteria:

* Patients with limited stage disease. This includes IA, IB, IIA, IIB, and IIIA.
* Age < 18 years old.
* History of a prior malignancy within three years with the exception of skin cancer (excluding melanoma), cervical carcinoma in situ, in situ breast carcinoma or stage A/B prostate cancer.
* Female patients who are pregnant or are breast feeding
* History of acute myocardial infarction or stroke within 6 months.
* Uncontrolled hypertension, unstable angina, New York Heart Association grade II or greater CHF, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease.
* Patients who have received other investigational drugs within 28 days.
* Patients with CNS involvement (brain or meningeal). The single exception to this is the patient previously treated for brain metastases with radiation therapy, or surgical excision who has no evidence of active residual metastases on brain MRI at the time of study entry.
* Patients with large neuroendocrine tumor or mixed small cell and non-small cell histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (16):
- United States (16):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Mercy Hospital, Portland, Maine
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Gandhi JG, Gian VG, Peyton JD, West-Osterfield K, Clark BL, Vazquez ER, Jones SF, Burris HA, Greco FA. A phase II trial of carboplatin and weekly topotecan in the first-line treatment of patients with extensive stage small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):862-6. doi: 10.1097/jto.0b013e3181d86a4f. PMID 20521352
- See also: Published article in the Journal of Thoracic Oncology — http://journals.lww.com/jto/pages/articleviewer.aspx?year=2010&issue=06000&article=00018&type=abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Topotecan/Carboplatin: Topotecan 4mg/m2 IV on days 1, 8. Carboplatin AUC=5 IV day 1 only . - Cycles are repeated every 21 days for > 4 cycles of topotecan and carboplatin (maximum 6 courses). Restaging studies will be performed every 2 cycles (or 6 weeks.)
Period: Overall Study
Arm/Group | Topotecan/Carboplatin
Started | 61
Completed | 23
Not Completed | 38

BASELINE CHARACTERISTICS:
Arm/Group | Topotecan/Carboplatin
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Overall response rate is the percent of patients experiencing a complete or partial response by RECIST v. 1 Criteria. Overall response rate is the percentage of patients with complete response or partial response per RECIST v.1 Criteria. Complete response (CR) = Disappearance of all target lesions, disappearance of all nontarget lesions for at least 4 weeks. Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
  The final response category assigned represented the best response obtained during treatment.
Time Frame: 18 months
Population: All patients were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Topotecan/Carboplatin
Number analyzed (Participants) | 61
percentage of participants | 57 [44 to 70]

2. Secondary Outcome: Time to Progression (TTP), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Time to progression is defined as the interval between the start date of treatment and the date of occurrence of progressive disease.
Time Frame: 18 months
Population: All patients were assessed for time to progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Topotecan/Carboplatin
Number analyzed (Participants) | 61
Months | 5.5 [4.0 to 6.3]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Overall survival was measured from the date of study entry until the date of death.
Time Frame: 18 months
Population: All patients were assessed for overall survival.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Topotecan/Carboplatin
Number analyzed (Participants) | 61
Months | 8.5 [7.2 to 11.4]

ADVERSE EVENTS:
Arm/Group | Topotecan/Carboplatin
Serious Adverse Events (participants affected / at risk) | 28/61
Other Adverse Events (participants affected / at risk) | 53/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan/Carboplatin (N=61)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conduction abnormality - Asystole (Cardiac disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Death not associated with CTCAE term - Disease Progression NOS (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Fever (NOS) (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal - Other (Gastroenteritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Perforated diverticulum) (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Hemorrhage, GI (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - Other (Cellulitis) (Infections and infestations) | 1 (1)
Infection - Other (Pneumonia) (Infections and infestations) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - chest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancytopenia (NOS) (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory Failure) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan/Carboplatin (N=61)
Alkaline Phospahatase (Metabolism and nutrition disorders) | 15 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (38)
ALT, SGPT (Metabolism and nutrition disorders) | 6 (9)
Anorexia (Gastrointestinal disorders) | 22 (50)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (19)
AST, SGOT (Metabolism and nutrition disorders) | 9 (11)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 16 (26)
Cardiac-Other (Cardiac disorders) | 4 (5)
Confusion (Nervous system disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 26 (70)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (27)
Dehydration (Gastrointestinal disorders) | 10 (18)
Diarrhea (Gastrointestinal disorders) | 16 (20)
Dizziness (Nervous system disorders) | 6 (10)
Dysphagia (Gastrointestinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (52)
Edema (Blood and lymphatic system disorders) | 11 (23)
Fatigue (General disorders) | 52 (184)
Febrile Neutropenia (Infections and infestations) | 6 (7)
Fever (General disorders) | 4 (5)
Hemoglobin (Blood and lymphatic system disorders) | 53 (200)
Hemorrhage (Lung) (Vascular disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (36)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (22)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 9 (10)
Hyponatremia (Metabolism and nutrition disorders) | 9 (11)
Hypotension (Cardiac disorders) | 8 (11)
Infection (Lung-Pneumonia) (Infections and infestations) | 6 (7)
Infection (Urinary Tract-NOS) (Infections and infestations) | 5 (6)
Insomnia (General disorders) | 11 (15)
Leukocytes (WBC) (Blood and lymphatic system disorders) | 46 (89)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 10 (12)
Mood Alteration (anxiety) (Nervous system disorders) | 6 (6)
Mood Alteration (Depression) (Nervous system disorders) | 8 (12)
Mucositis (Gastrointestinal disorders) | 5 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (12)
Nausea (Gastrointestinal disorders) | 26 (50)
Neutrophils (ANC/AGC) (Blood and lymphatic system disorders) | 53 (156)
Pain (General disorders) | 40 (96)
Pain (Abdomen-NOS) (Gastrointestinal disorders) | 6 (7)
Pain (back) (Musculoskeletal and connective tissue disorders) | 13 (19)
Pain (bone) (Musculoskeletal and connective tissue disorders) | 13 (27)
Pain (chest/thorax-NOS) (Respiratory, thoracic and mediastinal disorders) | 11 (20)
Pain (extremity-limb) (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain (headache) (Nervous system disorders) | 5 (5)
Pain (joint) (Musculoskeletal and connective tissue disorders) | 7 (11)
Pain (NOS) (General disorders) | 10 (13)
Platelets (Blood and lymphatic system disorders) | 50 (150)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 22 (41)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Sensory Neuropathy (Nervous system disorders) | 5 (10)
Skin (Skin and subcutaneous tissue disorders) | 12 (14)
Taste Alteration (Gastrointestinal disorders) | 4 (14)
Voice Changes/Dysarthria (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 16 (23)
Weight Loss (General disorders) | 12 (23)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.